CLINICAL TRIAL: NCT06738342
Title: Clinical Efficacy of a Chlorhexidine-based Mouth-rinse Containing Citrus Aurantium Amara in Patients Undergoing Periodontal Surgery: a Triple-blind, Parallel-arm, Randomized Controlled Trial
Brief Title: Clinical Efficacy of a Chlorhexidine-based Mouth-rinse Containing Citrus Aurantium Amara
Acronym: CUR_01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0460/2022
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: CHX 0.09% + Citrox + HA
- Control group (Active Comparator)
  Interventions: Drug: CHX 0.12%

INTERVENTIONS:
Other: CHX 0.09% + Citrox + HA — The patient will use the assigned mouthwash starting 24 hours after the surgical procedures and continuing twice a day for 14 days.
  Arms: Test group
Drug: CHX 0.12% — The patient will use the assigned mouthwash starting 24 hours after the surgical procedures and continuing twice a day for 14 days.
  Arms: Control group

SUMMARY:
The primary objective of the study is the evaluation of efficacy of a mouthwash cointaining Chlorexidine (CHX) 0.09% + HA + Citrox (test group) on the quality of wound healing and the presence plaque formation and gingival inflammation in the post-surgical phase. Futhermore stains, discolorations and adverse effects will be eventually recorded. Control group will be represented by the use of a CHX 0.12% mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* More than 20 natural teeth excluding the third molars
* Clinical indication for a surgical intervention for the treatment of at least one residual pocket after non-surgical therapy (pocket depth (PD) ≥5mm)
* Have a full mouth plaque score (FMPS) <15% before surgery;
* Have a full mouth bleeding score (FMBS) <15% before surgery;
* Ability and willingness to give written informed consent;
* Written agreement to participate in the trial.

Exclusion Criteria:

* Use of medications, such as anti-platelet or anti-coagulant agents, any other concomitant systemic disorder, cardiovascular and diabetes diseases, allergic, infectious diseases and medications affecting periodontal inflammation
* Pregnancy or breastfeeding;
* Use of medication affecting the healing process;
* Assumption of systemic or local antibiotics in the 4 weeks before trial beginning;
* Conditions of the teeth or of the site that contraindicate the surgery (severe mobility, fractures, untreated endodontic lesions, incongruous restorations);
* Patients with previous periodontal treatment or who were undergoing a course of dental or orthodontic treatment will be also excluded.
* Tobacco use (10 or more cigarettes per day)
* Inability to comply with protocol
* Uncooperative patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Oedema | 1, 3, 7 an 14 days
  Presence of absence will be recorded (1 or 0).

SECONDARY OUTCOMES:
Early Healing Score | 24 hours post surgery, 3, 7 and 45 days post surgery
  The score comprises three parameters (Clinical signs of re-epithelialization, hemostasis and inflammation) and ranges from 0 (worst healing) to 10 (best healing)
Plaque Index modified by Turesky | 1,3,7 and 14 days post surgery
Gingival Index modified by Trombelli | 1,3,7 and 14 days post surgery
Lobene Index modified | 1,3,7 and 14 days post surgery
  Presence of stains or discolorations of teeth and mucosae
Adverse effects | 1,3,7 and 14 days post surgery
  Disgeusia, mouth ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided